CLINICAL TRIAL: NCT00793104
Title: Evaluation of the Composite of Cancellous and Demineralized Bone Plug (CR-Plug) for Repair of Focal Cartilage Lesions in the Femoral Condyle
Brief Title: Evaluation of the CR Plug (Allograft) for the Treatment of a Cartilage Injury in the Knee.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrolment & potential regulatory changes for allograft in cartilage repair
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP2008; WIRB # 20081109 (Other: Western IRB); St Francis IRB Project # 571 (Other: St. Francis IRB)
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Knee Injury
Keywords: allograft; knee injury; cartilage injury; Osteochondral defects in the articular femoral cartilage
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CR Plug (Other): Placement of allograft CR Plug in primary injury site
  Interventions: Procedure: Placement of allograft CR Plug in primary injury site

INTERVENTIONS:
Procedure: Placement of allograft CR Plug in primary injury site — Core defect and implant allograft CR plug

SUMMARY:
Determine the ability of the allograft plug for the treatment of a cartilage injury in the knee

DETAILED DESCRIPTION:
The specific aim in this study is to assess the ability of the CR-Plug to treat osteochondral focal defects of less than 2.5 cm squared at high-load-bearing femoral condyle.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Skeletally mature
* Have one symptomatic score International Cartilage Repair Score (ICRS) grade 3a, 3b, 3c, 3d, 4a, 4b articular cartilage lesion less than 2.5 cm involving the Medial Femoral Condyle (MFC) or Lateral Femoral Condyle (LFC). Symptoms must include pain, pain with weight bearing and squatting, locking of joints, and/or swelling
* Functional meniscal tissue (defined as 5 mm or more width)
* A score of = or greater than 4 on the VAS questionnaire

Exclusion Criteria:

* Associated tibial or patellar articular cartilage defect greater than 2 ICRS
* Osteoarthritis of either knee
* Mechanical axis malalignment of greater than 5 degrees
* Patellofemoral incongruity of Merchant view
* One or more multiple defects greater than 2.5 cm
* Osteochondritis dissecans (OCD) with depth of bone loss greater than 4 mm
* Ligament treatments in the affected knee within one yer prior to current study
* Previous surgical meniscus treatments in the affected knee in the last 6 months
* Less than 5 mm of meniscal tissue in ipsilateral compartment of study treatment
* Use of any investigational therapy with in 30 days prior to the first visit
* Corticosteroid or viscosupplementation within the past 3 months
* A score of 3 or less on the VAS Questionnaire
* Active gout or pseudogout or systemic inflammatory condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Farr, MD, PhD, Principal Investigator — OrthoIndy, Inc; Ralph A Gambardella, MD, Principal Investigator — Kerlan Jobe Orthopaedic Clinic; Stewart Weinerman, MD, Principal Investigator — Colorado Orthopedic Consultants
Locations (3):
- United States (3):
  - Kerlan Jobe Orthopaedic Clinic, Los Angeles, California
  - Colorado Orthopedic Consultants, Denver, Colorado
  - OrthoIndy, Inc, Indianapolis, Indiana

REFERENCES:
- See also: Click here to find more information from OrthoIndy — http://www.orthoindy.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the patient population at two investigative sites between 17 November 2008 and 11 June 2010.
Pre-assignment Details: There was no group assignment
Period: Overall Study
Arm/Group | CR Plug
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | CR Plug
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Knee Injury and Osteoarthritis Outcome Score (KOOS) at 24 Months
Description: The outcome at 24 months as measured by the Knee injury and Osteoarthritis Outcome Score (KOOS). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Plug
Number analyzed (Participants) | 9
units on a scale | 86.04 (17.44)

2. Secondary Outcome: Current Health Assessment
Description: Evaluation on the Current Health Assessment at 24 months. Scores are transformed to a 0-100 scale, with zero representing a self-graded perception of extremely poor health and 100 representing no health problems. Scores between 0 and 100 represent the percentage of total possible score achieved.
Time Frame: 24 months, MRI only at 12 and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Plug
Number analyzed (Participants) | 9
units on a scale | 81.1 (22.0)

3. Secondary Outcome: Lysholm With Tegner Score
Description: The Tegner activity scale was designed as a score of activity level to complement other functional scores (eg the Lysholm knee score) for patients with ligamentous injuries. The instrument scores a person's activity level between 0 and 100 where 0 is 'on sick leave/disability' and 100 is 'participation in competitive sports at a full, unhindered level.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Plug
Number analyzed (Participants) | 9
units on a scale | 79.6 (22.0)

4. Secondary Outcome: International Knee Documentation Committee (IKDC) at 24 Months.
Description: The International Knee Documentation Committee scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Plug
Number analyzed (Participants) | 9
units on a scale | 79.4 (21.8)

5. Secondary Outcome: MRI Evaluation Score
Description: MRI images were graded by a radiologist with regard to the incorporation of the CR graft in both the cancellous and cortical portions of the bone at the graft site. The raw scores were converted to an index scale form 0 to 100, with 0 representing failure of the graft to incorporate and 100 representing complete incorporation of the graft.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Plug
Number analyzed (Participants) | 9
units on a scale | 95.5 (7.8)

ADVERSE EVENTS:
Arm/Group | CR Plug
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR Plug (N=10)
Graft Failure (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR Plug (N=10)
Mild knee effusion (Musculoskeletal and connective tissue disorders) | 10 (16)
Moderate knee effusion (Musculoskeletal and connective tissue disorders) | 4 (4)
reduced rom, KNEE (Musculoskeletal and connective tissue disorders) | 9 (9)
NAUSEA (Gastrointestinal disorders) | 4 (4)
whole body itching (General disorders) | 3 (3)
tingling sensation in foot (General disorders) | 1 (1)
knee catching (Musculoskeletal and connective tissue disorders) | 1 (1)
meniscus tear (Musculoskeletal and connective tissue disorders) | 1 (1)
plug protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
knee pain, mild (Musculoskeletal and connective tissue disorders) | 1 (1)
knee pain, moderate (Musculoskeletal and connective tissue disorders) | 1 (1)
knee pain after activity (Musculoskeletal and connective tissue disorders) | 1 (1)
increased knee pain, moderate (Musculoskeletal and connective tissue disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Enrollment was closed early due for 2 factors:

1) Slow enrollment and 2) A potential change in the regulatory pathway for allografts used in cartilage repair

1 patient was lost to follow up, with no data collected at the 24-month visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less